CLINICAL TRIAL: NCT04450030
Title: Immunoadsorption Versus High-dose Intravenous Corticosteroids in Relapsing Multiple Sclerosis - Assessment of Mechanism of Action
Brief Title: Immunoadsorption Versus High-dose Intravenous Corticosteroids in Relapsing Multiple Sclerosis
Acronym: INCIDENT-MS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Other Study IDs: INCIDENTMS2018
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-06

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: immunoadsorption; intravenous methyl prednisolone
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — methyl prednisolonate; Plasmapheresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intravenous methyl prednisolone: Patients receiving an additional course of intravenous methyl prednisolone for treatment of a steroid-refractory MS relapse
  Interventions: Drug: Methyl Prednisolonate
- Immunoadsorption: Patients receiving 6 courses of immunadsorption treatment for treatment of a steroid-refractory MS relapse
  Interventions: Procedure: Immunoadsorption

INTERVENTIONS:
Drug: Methyl Prednisolonate — 2000mg intravenous methyl prednisolone per day for five consecutive days
  Groups: Intravenous methyl prednisolone
Procedure: Immunoadsorption — 6 courses of tryptophane-based immunoadsorption within up to 12 days
  Groups: Immunoadsorption

SUMMARY:
Treatment of acute relapsing multiple sclerosis (MS) has remained largely unaltered within past years. However, evidence defining the exact role of apheresis treatment in the therapeutic sequence is still incomplete. INCIDENT-MS evaluates the mechanism of action of immunoadsorption compared to escalated methyl prednisolone treatment in steroid-refractory MS relapses and thereby will help to identify predictive markers for optimal treatment choice and will generate further insights into the pathophysiology of MS relapses.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Diagnosis of relapsing-remitting multiple sclerosis according to 2017 revised McDonald-criteria
* Incomplete remission of relapse symptoms following initiation treatment with 1000mg/d intravenous methyl prednisolone
* Absence of fever or clinically apparent signs of infection

Exclusion Criteria:

* Baseline EDSS score >6.5 points
* Previous administration of less than 3x1000mg or more than 5x1000mg IVMPS for initiation treatment
* Known pregnancy or rejection to perform a pregnancy test (female patients only)
* Immunosuppressive treatment for conditions other than multiple sclerosis
* Ongoing neoplastic disorder or past neoplastic disorder within previous five years
* Known or newly diagnosed HIV-, HBV- or HCV-infection
* Regular intake of ACE inhibitor drugs
* Known bleeding disorders (including laboratory abnormalities such as: (I) platelet count<50.000/µL; (II) international normalized ratio>1.5, (III) activated prothrombin time>50s) or intake of oral anticoagulant drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute relapsing multiple sclerosis that were refractory to a first course of intravenous methyl prednisolone (1000mg per day for three to five consecutive days)
Sampling Method: Probability Sample
Enrollment: 204 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-09-05 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Expanded disability status scale (EDSS) | 2 weeks
  Improvement of disability compared to peak relapse EDSS following escalation treatment compared to peark relapse values

SECONDARY OUTCOMES:
visual-evoked potentials (VEP; P100-latency) | 2 weeks; 6 to 8 weeks
  Evolution of VEP P100-latency compared to peak relapse values
somatosensory-evoked potentials (SEP; Medianus and Tibialis; N20-, P40-latency) | 2 weeks; 6 to 8 weeks
  Evolution of SEP N20-/P40-latency compared to peak relapse values
best-corrected visual acuity (bcVA) | 2 weeks; 6 to 8 weeks
  Evolution of bcVA compared to peak relapse values
Expanded disability status scale (EDSS) | 6 to 8 weeks
  Confirmation of improvement of disability compared to primary endpoint
Multiple scleroris functional compositie (MSFC) | 2 weeks, 6 to 8 weeks
  Development of MSFC z-score compared to peak relapse values
Short form-36 questionaire (SF-36) | 6 to 8 weeks
  Development of quality-of-life compared to peak relapse values

CONTACTS AND LOCATIONS:
Overall Officials: Sven G Meuth, Prof Dr, Principal Investigator — University Hospital Muenster, Department of Neurology
Locations (1):
- Department of Neurology with Institute of Translational Neurology, University Hospital Muenster, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pfeuffer S, Rolfes L, Wirth T, Steffen F, Pawlitzki M, Schulte-Mecklenbeck A, Gross CC, Brand M, Bittner S, Ruck T, Klotz L, Wiendl H, Meuth SG. Immunoadsorption versus double-dose methylprednisolone in refractory multiple sclerosis relapses. J Neuroinflammation. 2022 Sep 7;19(1):220. doi: 10.1186/s12974-022-02583-y. PMID 36071461